CLINICAL TRIAL: NCT01485796
Title: Tolerability, Safety and Administration Mode Evaluation of Recombinant Human Hyaluronidase (rHuPH20) Facilitated Subcutaneous Treatment With Immune Globulin Infusion (Human), 10% in Subjects With Primary Immunodeficiency Diseases (PIDD)
Brief Title: Tolerability and Safety of IGI, 10% With rHuPH20 in PIDD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161101
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: PIDD
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epoch 1 and Epoch 2 (Experimental): In Study Epoch 1 PIDD patients that are already on intravenous treatment or subcutaneous treatment will be enrolled and treated with IGI, 10% and rHuPH20 subcutaneously, with a short dose/interval ramp-up (Epoch 1) consisting of one 1-week dose and interval and one 2-week dose and interval. The ramp-up (Epoch 1) is followed by Epoch 2 which consists of approximately 6 months (24 weeks) of IGI, 10% and rHuPH20 treatment. For subjects pretreated intravenously (IV), this treatment will occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), depending on the subject´s previous IV dosing schedule. For subjects pretreated subcutaneously (SC), treatment will also occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), at the discretion of the investigator and subject.
  Interventions: Biological: Immune Globulin Infusion (Human), 10%; Biological: Recombinant human hyaluronidase

INTERVENTIONS:
Biological: Immune Globulin Infusion (Human), 10% — Subcutaneous administration will be used in Study Epochs 1 and 2.
  Other Names: IGI; 10%
Biological: Recombinant human hyaluronidase — rHuPH20 will be administered subcutaneously (SC) immediately before each SC IGI, 10% infusion, through the same needle, at a rate of 1 to 2 mL/min.
  Other Names: rHuPH20

SUMMARY:
The purpose of the study is to acquire additional data on safety and tolerability of recombinant human hyaluronidase (rHuPH20) facilitated subcutaneous treatment of Immune Globulin Infusion (Human), 10% (IGI, 10%) and to assess the mode of product administration.

Following a discussion with the FDA at the end of July 2012, all participants still active in the study stopped treatment with rHuPH20 to assure safety of the participants participating in the study and went into a safety follow-up.

During this safety follow-up period, participants underwent treatment with the licensed product IGI, 10% (Gammagard Liquid). The intravenous or subcutaneous administration route was at the discretion of the participant and the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of a form of primary humoral immunodeficiency involving a defect in antibody formation and requiring gammaglobulin replacement, as defined according to the IUIS Scientific Committee 2009 and by diagnostic criteria according to Conley et al. The diagnosis must be reviewed by the Medical Director prior to enrollment.
* Subject is 2 years or older at the time of screening.
* Written informed consent is obtained from either the subject or the subject's legally authorized representative prior to any study-related procedures and study product administration.
* Subject has been receiving a consistent dose of immunoglobulin G (IgG) with a non-Baxter product (Gammunex administered IV, Hizentra, or Privigen), administered in compliance with the respective product information, for a period of at least 3 months prior to screening. The average minimum pre-study dose over that interval was equivalent to 300 mg/kg BW/4 weeks and a maximum dose equivalent to 600 mg/kg BW/4 weeks at a dosing frequency as follows:

  * For IV treatment prior to the study: at mean intervals of 3 or 4 weeks (+/- 3 days) or
  * For SC treatment prior to the study: at mean intervals of approximately 1 or 2 weeks (+/- 2 days).
* Subject has a serum trough level of IgG > 5 g/L at screening.
* Subject has not had a serious bacterial infection within the 3 months prior to screening.
* If female of childbearing potential, subject presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
* Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Subject has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2.
* Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

  * Persistent alanine aminotransferase (ALT) and aspartate amino transferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
  * Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] <= 500/mm3).
* Subject has creatinine clearance (CLcr) value that is <60% of normal for age and gender either measured, or calculated according to a gender-specific formula provided in the study protocol.
* Subject has been diagnosed with or has a malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix), unless the disease-free period prior to screening exceeds 5 years
* Subject is receiving anti-coagulation therapy or has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) within 12 months prior to screening or a history of thrombophilia.
* Subject has abnormal protein loss (protein losing enteropathy, nephrotic syndrome).
* Subject has anemia that would preclude phlebotomy for laboratory studies, according to standard practice at the site.
* Subject has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IV immunoglobulin, SC immunoglobulin, and/or Immune Serum Globulin (ISG) infusions.
* Subject has immunoglobulin A (IgA) deficiency (IgA less than 0.07g/L) and known anti IgA antibodies.
* Subject has a known allergy to hyaluronidase.
* Subject is on preventative (prophylactic) systemic antibacterial antibiotics at doses sufficient to treat or prevent bacterial infections, and cannot stop these antibiotics at the time of screening.
* Subject has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening.
* Subject has a bleeding disorder or a platelet count less than 20,000/μL, or who, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of SC therapy.
* Subject has total protein > 9 g/dL or myeloma, or macroglobulinemia (IgM) or paraproteinemia.
* Women of childbearing potential meeting any one of the following criteria:

  * Subject presents with a positive pregnancy test
  * Subject is breast feeding
  * Subject intends to begin nursing during the course of the study
  * Subject does not agree to employ adequate birth-control measures (e.g. intrauterine device, diaphragm or condom [for male partner] with spermicidal jelly or foam, or birth control pills/patches) throughout the course of the study.
* Subject has participated in another clinical study and has been exposed to an investigational product (IP) or device within 30 days prior to study enrollment (exception: treatment with immunoglobulin pre-study).
* Subject is scheduled to participate in another (non-Baxter) clinical study involving an IP or device during the course of the study.
* Subject has severe dermatitis that would preclude adequate sites for safe product administration.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (10):
  - University of California, Irvine, Irvine, California
  - IMMUNOe International Research Centers, Thornton, Colorado
  - Allergy Associates of the Palm Beaches, PA, North Palm Beach, Florida
  - LSU Health Sciences Center & Children´s Hospital, New Orleans, Louisiana
  - Midwest Immunology, Plymouth, Minnesota
  - Midlands Pediatrics PC, Papillion, Nebraska
  - Winthrop Allergy and Immunology, Mineola, New York
  - Oklahoma Institute of Allergy & Asthma Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Allergy, Asthma & Immunology Clinic PA, Irving, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 16 study sites in the US.
Pre-assignment Details: Of 54 subjects screened for the study, 37 started treatment. Of the 17 subjects who discontinued the study before treatment, 10 were screen failures, 5 withdrew consent, and for 2 subjects enrollment ended due to other reasons.
Groups:
- Subcutaneous Treatment With IGI, 10% and rHuPH20: Subcutaneous treatment with IGI, 10% and rHuPH20 occurred in 2 study epochs. In Epoch 1, PIDD patients that were already on intravenous (IV) or subcutaneous (SC) treatment were treated with IGI, 10% and rHuPH20 subcutaneously, with one 1-week dose and interval and one 2-week dose and interval. Epoch 2 was to consist of approx. 6 months (24 weeks) of IGI, 10% and rHuPH20 treatment. For subjects pretreated IV, this treatment was to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), depending on the subject´s previous IV dosing schedule. For subjects pretreated SC, treatment was also to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), at the discretion of the investigator and subject. However, treatment with rHuPH20 was stopped as of August 2012 following a discussion with the FDA, and subjects still active in Epoch 2 were switched to a safety follow-up. During the safety-follow up, subjects received IGI, 10% by either the IV or the SC route.
Period: Period 1: Epoch 1 (Ramp-up)
Arm/Group | Subcutaneous Treatment With IGI, 10% and rHuPH20
Started | 37
Treated in Epoch 1 | 37
Completed | 36
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2: Epoch 2
Arm/Group | Subcutaneous Treatment With IGI, 10% and rHuPH20
Started | 36
Treated in Epoch 2 | 36
Completed | 1
Not Completed | 35
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 3
Not completed — Switch to safety follow-up | 26
Period: Overall Trial (Incl. Safety Follow-up)
Arm/Group | Subcutaneous Treatment With IGI, 10% and rHuPH20
Started | 37
Treated in Epoch 1 (Ramp-up) | 37
Completed Epoch 1 (Ramp-up) | 36
Started Epoch 2 | 36
Treated in Epoch 2 | 36
Completed Epoch 2 | 1
Switch to Safety Follow-up | 26
Completed Safety Follow-up | 24
Completed | 25 (1 subject who completed Epoch 2 + 24 subjects who completed the safety follow-up)
Not Completed | 12
Not completed — Withdrawal by Subject in Epoch 1 | 1
Not completed — Withdrawal by Subject in Epoch 2 | 6
Not completed — Adverse Event in Epoch 2 | 3
Not completed — Withdrawal During Safety-Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Subcutaneous Treatment With IGI, 10% and rHuPH20: This analysis set comprises all subjects exposed to study drug in Epoch 1 and Epoch 2. In Epoch 1, PIDD patients that were already on intravenous (IV) or subcutaneous (SC) treatment were treated with IGI, 10% and rHuPH20 subcutaneously, with one 1-week dose and interval and one 2-week dose and interval. Epoch 2 was to consist of approx. 6 months (24 weeks) of IGI, 10% and rHuPH20 treatment. For subjects pretreated IV, this treatment was to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), depending on the subject´s previous IV dosing schedule. For subjects pretreated SC, treatment was also to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), at the discretion of the investigator and subject. However, treatment with rHuPH20 was stopped as of August 2012 following a discussion with the FDA, and subjects still active in Epoch 2 were switched to a safety follow-up (IGI, 10% by IV or SC route).
Arm/Group | Subcutaneous Treatment With IGI, 10% and rHuPH20
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: Years] | 33.0 [6 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Related Systemic Adverse Events (Excluding Infections)
Time Frame: 7 months (per subject)
Measure: Number; unit: adverse events
Groups:
- Safety Analysis Set (n=37): The Safety Analysis Set comprises all subjects exposed to study drug in Epoch 1 and Epoch 2.
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
adverse events | 59

2. Primary Outcome: Rate of Related Systemic Adverse Events (Excluding Infections) Per Infusion
Description: A point estimate and 95% confidence interval for the rate of related systemic adverse events per infusion was derived using a Poisson model.
Time Frame: 7 months (per subject)
Measure: Number (95% Confidence Interval); unit: adverse events
Groups:
- Epoch 2 Data Set (n=36): The Epoch 2 Data Set comprises all subjects of the safety analysis set who received study drug in Epoch 2.
Arm/Group | Safety Analysis Set (n=37) | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 37 | 36
adverse events
  Epoch 1 | 0.250 [0.140 to 0.406] | 0.253 [0.141 to 0.413]
  Epoch 2 | 0.377 [0.205 to 0.626] | 0.377 [0.205 to 0.626]
  Epoch 1+2 | 0.324 [0.187 to 0.517] | 0.326 [0.186 to 0.522]

3. Secondary Outcome: Proportion of Subjects Who Achieve a Treatment Interval of 3 or 4 Weeks in Epoch 2
Time Frame: 6 months (per subject)
Measure: Number; unit: subjects
Arm/Group | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 36
subjects
  3 or 4-week treatment interval | 36
  3-week treatment interval | 6
  4-week treatment interval | 30

4. Secondary Outcome: Proportion of Subjects Who Maintain a Treatment Interval of 3 or 4 Weeks in Epoch 2 for 24 Weeks
Time Frame: 6 months (per subject)
Measure: Number; unit: subjects
Arm/Group | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 36
subjects | 1

5. Secondary Outcome: Number of Related Local Adverse Events (Excluding Infections)
Time Frame: 7 months (per subject)
Measure: Number; unit: adverse events
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
adverse events | 153

6. Secondary Outcome: Rate of Related Local Adverse Events (Excluding Infections) Per Infusion
Description: A point estimate and 95% confidence interval for the rate of related local adverse events per infusion was derived using a Poisson model.
Time Frame: 7 months (per subject)
Measure: Number (95% Confidence Interval); unit: adverse events
Arm/Group | Safety Analysis Set (n=37) | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 37 | 36
adverse events
  Epoch 1 | 0.882 [0.581 to 1.271] | 0.880 [0.575 to 1.278]
  Epoch 2 | 0.811 [0.541 to 1.160] | 0.811 [0.541 to 1.160]
  Epoch 1+2 | 0.841 [0.587 to 1.159] | 0.840 [0.582 to 1.164]

7. Secondary Outcome: Number of All Related Adverse Events (Excluding Infections)
Time Frame: 7 months (per subject)
Measure: Number; unit: adverse events
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
adverse events | 212

8. Secondary Outcome: Rate of All Adverse Events (Excluding Infections) Per Infusion
Description: A point estimate and 95% confidence interval for the rate of adverse events per infusion was derived using a Poisson model.
Time Frame: 7 months (per subject)
Measure: Number (95% Confidence Interval); unit: adverse events
Arm/Group | Safety Analysis Set (n=37) | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 37 | 36
adverse events
  Epoch 1 | 1.645 [1.221 to 2.157] | 1.653 [1.221 to 2.178]
  Epoch 2 | 1.642 [1.164 to 2.235] | 1.642 [1.164 to 2.235]
  Epoch 1+2 | 1.643 [1.235 to 2.132] | 1.646 [1.232 to 2.145]

9. Secondary Outcome: Number of Subjects Who Develop Neutralizing Antibodies to rHuPH20
Time Frame: 7 months (per subject)
Measure: Number; unit: subjects
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
subjects | 0

10. Secondary Outcome: Trough Levels of Immunoglobulin G (IgG)
Description: IgG trough levels at the beginning of Study Epoch 1 (previous immunoglobulin treatment) and at the end of Study Epoch 2 were analyzed.
Time Frame: 7 months (per subject)
Population: At screening, data (ie, IgG trough levels) were available for analysis from 36 participants. At the end of Epoch 2, data were available for analysis from only 33 participants.
Measure: Geometric Mean (95% Confidence Interval); unit: g/L
Groups:
- Epoch 2 Data Set: The Epoch 2 Data Set comprises all subjects of the safety analysis set who received study drug in Epoch 2.
Arm/Group | Epoch 2 Data Set
Number analyzed (Participants) | 36
g/L
  At screening | 10.53 [9.46 to 11.73]
  At end of Epoch 2: number analyzed (Participants) | 33
  At end of Epoch 2 | 9.21 [8.28 to 10.25]

11. Secondary Outcome: Number of Infusions Per Month in Epoch 1 and Epoch 2
Description: Non-parametric descriptive statistics (median, range) are provided.
Time Frame: 7 months (per subject)
Population: The number of participants analyzed for Epoch 1 is 37, as 37 participants were treated with study drug in Epoch 1. The number of participants analyzed for Epoch 2 is 36, as 36 participants were treated with study drug in Epoch 2.
Measure: Median (Full Range); unit: infusions
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
infusions
  Epoch 1 | 2.90 [2.5 to 10.1]
  Epoch 2: number analyzed (Participants) | 36
  Epoch 2 | 1.09 [0.6 to 2.0]

12. Secondary Outcome: Number of Infusion Sites (Needle Sticks) Per Month in Epoch 1 and Epoch 2
Description: Non-parametric descriptive statistics (median, range) are provided.
Time Frame: 7 months (per subject)
Population: as for outcome 11
Measure: Median (Full Range); unit: infusion sites (needle sticks)
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
infusion sites (needle sticks)
  Epoch 1 | 2.90 [2.5 to 10.1]
  Epoch 2: number analyzed (Participants) | 36
  Epoch 2 | 1.12 [0.6 to 3.8]

13. Secondary Outcome: Duration of Infusion in Epoch 1 and Epoch 2
Description: Non-parametric descriptive statistics (median, range) are provided.
Time Frame: 7 months (per subject)
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
hours
  Epoch 1 | 1.23 [0.53 to 3.10]
  Epoch 2: number analyzed (Participants) | 36
  Epoch 2 | 1.67 [0.80 to 3.55]

14. Secondary Outcome: Maximum Infusion Rate in Epoch 1 and Epoch 2
Description: Non-parametric descriptive statistics (median, range) are provided.
Time Frame: 7 months (per subject)
Population: as for outcome 11
Measure: Median (Full Range); unit: mL/h
Arm/Group | Safety Analysis Set (n=37)
Number analyzed (Participants) | 37
mL/h
  Epoch 1 | 240.0 [60 to 300]
  Epoch 2: number analyzed (Participants) | 36
  Epoch 2 | 300.0 [10 to 300]

15. Secondary Outcome: Number of Weeks to Reach Final 3 or 4-week Dose Interval
Description: Non-parametric descriptive statistics (median, range) are provided.
Time Frame: 7 months (per subject)
Population: Of 36 participants treated with study drug in Epoch 2, 6 reached a final dose interval of 3 weeks and 30 reached a final dose interval of 4 weeks.
Measure: Median (Full Range); unit: weeks
Arm/Group | Epoch 2 Data Set (n=36)
Number analyzed (Participants) | 36
weeks
  3-week dose interval: number analyzed (Participants) | 6
  3-week dose interval | 3.0 [3 to 5]
  4-week dose interval: number analyzed (Participants) | 30
  4-week dose interval | 3.0 [3 to 4]

ADVERSE EVENTS:
Time Frame: Overall: Approximately 1 year Per subject: 7 months
Groups:
- Epochs 1+2 (SC Treatment w/ IGI,10% and rHuPH20, n=37): This analysis set comprises all subjects exposed to study drug in Epoch 1 and Epoch 2. In Epoch 1, PIDD patients that were already on intravenous (IV) or subcutaneous (SC) treatment were treated with IGI, 10% and rHuPH20 subcutaneously, with one 1-week dose and interval and one 2-week dose and interval. Epoch 2 was to consist of approx. 6 months (24 weeks) of IGI, 10% and rHuPH20 treatment. For subjects pretreated IV, this treatment was to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), depending on the subject´s previous IV dosing schedule. For subjects pretreated SC, treatment was also to occur every 3 or 4 weeks (at a 3-week or 4-week dose, respectively), at the discretion of the investigator and subject. However, treatment with rHuPH20 was stopped as of August 2012 following a discussion with the FDA, and subjects still active in Epoch 2 were switched to a safety follow-up (IGI, 10% by IV or SC route).
- Safety Follow-up (n=26): Treatment with rHuPH20 was stopped as of August 2012 following discussion with the FDA. This decision was based on theoretical risks of exposure to anti-rHuPH20 antibodies, not because of any clinical adverse events. 26 subjects still active in Epoch 2 of the study went into a safety follow-up period and were treated with IGI, 10% (GAMMAGARD LIQUID) either intravenously or subcutaneously.
Arm/Group | Epochs 1+2 (SC Treatment w/ IGI,10% and rHuPH20, n=37) | Safety Follow-up (n=26)
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/26
Other Adverse Events (participants affected / at risk) | 30/37 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epochs 1+2 (SC Treatment w/ IGI,10% and rHuPH20, n=37) (N=37) | Safety Follow-up (n=26) (N=26)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — This event occurred during the safety follow-up period. It was resolved by the time of study completion.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epochs 1+2 (SC Treatment w/ IGI,10% and rHuPH20, n=37) (N=37) | Safety Follow-up (n=26) (N=26)
Upper abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (10) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (6) | 0 (0)
Infusion site discoloration (General disorders) | 4 (11) | 0 (0)
Infusion site erythema (General disorders) | 11 (26) | 0 (0)
Infusion site hematoma (General disorders) | 2 (2) | 0 (0)
Infusion site pain (General disorders) | 21 (64) | 0 (0)
Infusion site pruritus (General disorders) | 5 (8) | 0 (0)
Infusion site swelling (General disorders) | 9 (23) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Local swelling (General disorders) | 4 (9) | 0 (0)
Pain (General disorders) | 3 (4) | 1 (2)
Pyrexia (General disorders) | 5 (6) | 2 (4)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 10 (25) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Hemosiderinuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Treatment with rHuPH20 was stopped as of August 2012 following discussion with the FDA. 26 subjects still active in Study Epoch 2 went into a safety follow-up period and were treated with IGI, 10% (GAMMAGARD LIQUID) intravenously or subcutaneously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxalta requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxalta may request an additional delay of ≤60 days eg, for intellectual property protection.